CLINICAL TRIAL: NCT04689490
Title: Prospective Study of Persistent Dyspnea in Recovered COVID-19 Patients
Acronym: DISCOVID19
Status: Completed | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Ignacio J. Amat Santos, Coordinator of Interventional Cardiology Unit, Hospital Clínico Universitario de Valladolid
Other Study IDs: CASVE PI-20-1894
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Dyspnea
Keywords: Dyspnea; Covid19; Cardiopulmonary exercise test
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Exercise Test; Respiratory Function Tests; Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dyspnea: Patients with prior hospitalization because of COVID-19, with succesful hospital discharge, who underwent at least a first-time follow-up from the index event, and present persistent dyspnea.
  Interventions: Diagnostic Test: Cardiopulmonary exercise test
- Control: Patients with prior hospitalization because of COVID-19, with succesful hospital discharge, who underwent at least a first-time follow-up from the index event, fully recovered, without persistent dyspnea.
  Interventions: Diagnostic Test: Cardiopulmonary exercise test

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test — Only diagnostic tests
  Other Names: walking test; pulmonary lung test; echocardiography; blood sampling

SUMMARY:
We conducted a national, single center (Hospital Clínico Universitario de Valladolid, Spain, Valladolid), prospective study of patients with prior hospitalization because of COVID-19 who were admitted between March 1st, 2020, and May 15th, 2020. All eligible patients underwent at least at first-time follow-up from the index event. Exclusion criteria were age < 18 years old, pregnant women, terminally ill patients, active SARS-CoV-2 infections, inability to exercise and previous known severe pulmonary or heart disease. Patients underwent a clinical assessment for symptom burden, questionnaire for quality of life (Kansas City Cardiomyopathy Questionnaire and SF-36), venous blood sampling, 6-minute walking test (6-MWT), tests of lung function (spirometry and diffusing capacity of the lungs for carbon monoxide) and treadmill cardio-pulmonary exercise testing (CPET). 48-hours before the test of lung function and the CPET, all patients yielded a negative result in the reverse transcription-polymerase chain reaction (RT-PCR) for SARS-CoV-2. For definitive analysis patients were assigned to the control group if they did not refer dyspnea at the time of the follow-up, a small asymptomatic out-patient control group without prior hospitalization was also included.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Previous COVID-19 hospitalization with successful discharged
* Availability of at least one follow up per clinical protocol

Exclusion Criteria:

* pregnant women
* terminally ill patients
* active SARS-CoV-2 infections
* inability to exercise
* previous known severe pulmonary or heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with prior hospitalization because of COVID-19 who were admitted between March and May. All eligible patient underwent at least at first-time follow-up from the index event. Exclusion criteria were age < 18 years old, pregnant women, terminally ill patients, active SARS-CoV-2 infections, inability to exercise and previous known severe pulmonary or heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity | 6 months
  Measured as peak oxygen uptake
Total Lung Capacity (TLC) | 6 months
  Pulmonary function test
Force Expiratory Volume in 1 second (FEV1) | 6 months
  Pulmonary function test
Difussing Lung Capacity of CO (DLCO) | 6 months
  Pulmonary function test
Forced Vital Capacity (FVC) | 6 months
  Pulmonary function test
Left Ventricular (LV) Function | 6 months
  Left Ventricular (LV) Function (Ecocardiagraphy-measured Cardiac Function)
Right Ventricular (RV) Function | 6 months
  Right Ventricular (RV) Function (Ecocardiagraphy-measured Cardiac Function)

SECONDARY OUTCOMES:
Short Form 36 Health Survey (SF-36) | 6 months
  Quality of Life test
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 Months
  Quality of Life test
6 Minute Walk Test | 6 months
  Walking capacity
N-terminal pro hormone B-type natriuretic peptide (NT-proBNP) | 6 months
  Inflammatory and Cardiac Marker
Troponin-T | 6 months
  Inflammatory and Cardiac Marker
Ferritin | 6 months
  Inflammatory and Cardiac Marker
D-Dimer | 6 months
  Inflammatory and Cardiac Marker
interleukine-6 | 6 months
  Inflammatory and Cardiac Marker
C reactive protein (CRP) | 6 months
  Inflammatory and Cardiac Marker

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinney SP, Giustino G, Halperin JL, Mechanick JI, Neibart E, Olin JW, Rosenson RS, Fuster V. Coronavirus Historical Perspective, Disease Mechanisms, and Clinical Outcomes: JACC Focus Seminar. J Am Coll Cardiol. 2020 Oct 27;76(17):1999-2010. doi: 10.1016/j.jacc.2020.08.058. PMID 33092736
- [Background] Ahmed H, Patel K, Greenwood DC, Halpin S, Lewthwaite P, Salawu A, Eyre L, Breen A, O'Connor R, Jones A, Sivan M. Long-term clinical outcomes in survivors of severe acute respiratory syndrome and Middle East respiratory syndrome coronavirus outbreaks after hospitalisation or ICU admission: A systematic review and meta-analysis. J Rehabil Med. 2020 May 31;52(5):jrm00063. doi: 10.2340/16501977-2694. PMID 32449782
- [Result] Aparisi A, Ybarra-Falcon C, Garcia-Gomez M, Tobar J, Iglesias-Echeverria C, Jaurrieta-Largo S, Ladron R, Uribarri A, Catala P, Hinojosa W, Marcos-Mangas M, Fernandez-Prieto L, Sedano-Gutierrez R, Cusacovich I, Andaluz-Ojeda D, de Vega-Sanchez B, Recio-Platero A, Sanz-Patino E, Calvo D, Baladron C, Carrasco-Moraleja M, Disdier-Vicente C, Amat-Santos IJ, San Roman JA. Exercise Ventilatory Inefficiency in Post-COVID-19 Syndrome: Insights from a Prospective Evaluation. J Clin Med. 2021 Jun 11;10(12):2591. doi: 10.3390/jcm10122591. PMID 34208271